CLINICAL TRIAL: NCT02518412
Title: Transcranial Direct Current Stimulation (tDCS) as a Cognitive Enhancer for Patients With Alzheimers Disease
Acronym: tDCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012/1890(REK)
Record Dates: First submitted 2015-06-08; First posted 2015-08-07 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Alzheimer Disease
Keywords: Alzheimers disease; Transcranial direct current stimulation (tDCS); Neuromodulation; Neuropsychology
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active tDCS (Experimental): Participants receive active tDCS stimulation. Half of the participants receive active tDCS stimulation, i.e 30 minutes active stimulation of the temporal cortex.
  Interventions: Other: tDCS
- Placebo tDCS (Placebo Comparator): Participants receive placebo tDCS stimulation. Half of the participants receive placebo tDCS stimulation, i.e 30 minutes inactive stimulation of the temporal cortex.
  Interventions: Other: Placebo tDCS

INTERVENTIONS:
Other: tDCS — Transcranial Direct Current Stimulation (tDCS) is a non-invasive treatment method, using a low Direct current stimulation to increase excitability and thus stimulate plasticity and cognitive functions.
  Arms: Active tDCS
Other: Placebo tDCS — Half of the patients will receive Placebo tDCS. The procedure is the same as for active tDCS, but the in the Placebo tDCS the stimulation is non-active / sham.
  Arms: Placebo tDCS

SUMMARY:
The purpose of this study is to investigate transcranial direct current stimulation (tDCS) as a cognitive enhancer for patients with Alzheimer disease.

Transcranial direct current stimulation (tDCS) is a neuromodulation technique, that are applied to the brain by using two electrodes. These electrodes are placed on the scalp. The current is low intensity, usually 1-2 milliampere. tDCS may affect cognitive functions by increasing cortical excitability. tDCS is regarded as a safe treatment approach. In the present study, participants will undergo six stimulations. The effect of all stimulations swill be measured with neuropsychological testing before the first (pre) and after the sixth tDCS stimulation (post).

DETAILED DESCRIPTION:
The present study is a randomized controlled study (RCT) and will use tDCS to stimulate left temporal lobe and hopefully improve verbal memory functions. A total of 30 patients with Alzheimer disease will receive tDCS treatment for 30 minutes, six times. Half of the patients will undergo sham stimulation. These six stimulations will be executed during 10 days. Patients will be tested with neuropsychological tests before the first stimulation and after the last stimulation to assess the effect of the treatment. Patients will be retested six months later in order to investigate long-term effects ot the stimulation. The main hypothesis in the present study is that tDCS stimulation will lead to significant improvements in verbal memory functions.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimers disease according to (National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association).
* The cognitive impairment and decline must be documented by cognitive / neuropsychological testing and from an informant.

Exclusion Criteria:

* Stroke,
* Cancer,
* Psychiatric disorders (major depression, psychosis) or diseases / injuries in the central nervous system.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological testing | Changes in results from neuropsychological testing pre (before the first stimulation) og post treatment (after the last stimulation). There will be a ten days time frame from pre-test to post-test.
  We will use a neuropsychological test called California Verbal Learning Test and test verbal memory functions before the first treatment session and after the last treatment session. We will use this test to assess how the tDCS intervention will affect verbal memory functions. There will be a maximum of ten days between pre and post testing, since the entire stimulation procedure (six stimulations) will be executed during ten days.

CONTACTS AND LOCATIONS:
Overall Officials: Per M Aslaksen, PhD, Study Director — University of Tromso
Locations (1):
- Department of Psychology, University of Tromsø, Tromsø, Norway

REFERENCES:
- [Derived] Bystad M, Gronli O, Rasmussen ID, Gundersen N, Nordvang L, Wang-Iversen H, Aslaksen PM. Transcranial direct current stimulation as a memory enhancer in patients with Alzheimer's disease: a randomized, placebo-controlled trial. Alzheimers Res Ther. 2016 Mar 23;8(1):13. doi: 10.1186/s13195-016-0180-3. PMID 27005937